CLINICAL TRIAL: NCT02344758
Title: Non-invasive Gluten-free Diet Adherence Monitoring in Celiac Patients: Detection of Gluten Immunogenic Peptides in Urine
Brief Title: Gluten-free Diet Monitoring in Urine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Instituto Hispalense de Pediatría (Unknown); Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Carolina Sousa Martin, Professor, University of Seville
Allocation: Randomized | Model: Parallel
Other Study IDs: CELIFLUID1
Record Dates: First submitted 2015-01-14; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Celiac adult (Experimental): Patient >16 years, initially diagnosed based on the detection of IgA anti-endomysial and anti-tissue transglutaminase antibodies in serum and confirmed by a small intestinal biopsy, on a GFD for >2 years
  Interventions: Device: Non-invasive lateral flow test for monitoring gluten intake; Behavioral: gluten-free diet (GFD)
- Celiac child (Experimental): Patient <16 years, initially diagnosed based on the detection of IgA anti-endomysial and anti-tissue transglutaminase antibodies in serum and confirmed by a small intestinal biopsy, on a GFD for >2 years
  Interventions: Device: Non-invasive lateral flow test for monitoring gluten intake; Behavioral: gluten-free diet (GFD)
- Healthy adult (Active Comparator): Healthy individual > 16 years. Exclusion criteria: the presence of family history of CD, digestive disease symptoms, known medical disease, use of prescription medications, and use of antibiotics and probiotics in the previous 2 months to the inclusion in the study.
  Interventions: Device: Non-invasive lateral flow test for monitoring gluten intake; Behavioral: gluten-containing diet
- Healthy child (Active Comparator): Healthy individual < 16 years. Exclusion criteria: the presence of family history of CD, digestive disease symptoms, known medical disease, use of prescription medications, and use of antibiotics and probiotics in the previous 2 months to the inclusion in the study.
  Interventions: Device: Non-invasive lateral flow test for monitoring gluten intake; Behavioral: gluten-containing diet

INTERVENTIONS:
Device: Non-invasive lateral flow test for monitoring gluten intake
Behavioral: gluten-free diet (GFD)
  Arms: Celiac adult; Celiac child
Behavioral: gluten-containing diet
  Arms: Healthy adult; Healthy child

SUMMARY:
The purpose of this study is to develope a novel method to determine gluten intake and to check gluten-free diet adherence in celiac patients by detection of gluten immunogenic peptides in urine.

DETAILED DESCRIPTION:
To date, the mainstay of the management of CD is a strict life-long adherence to gluten-free diet (GFD). Follow-up monitoring of the improvement of patients on GFD is essential to assess symptomatic recovery and to monitor complications, as well as to assist patients with dietary compliance. However, practical methods to monitor diet compliance and to detect the origin of an outbreak of celiac clinical symptoms are not available.

In this study, we have overcome these challenges and shown the feasibility of measuring gluten immunogenic peptides (GIP) in urine samples in healthy and celiac individuals by solid phase extraction and estimating the peptide concentrations with a reader of anti-GIP moAb immunochromatographic strips (IC-strips).

ELIGIBILITY:
Inclusion Criteria:

* Celiac patient: childs (< 16 years) and adults (> 16 years)
* written informed consent

Exclusion Criteria:

* presence of family history of CD
* digestive disease symptoms
* known medical disease
* use of prescription medications and use of antibiotics and probiotics in the previous 2 months to the inclusion in the study
* participation in any other studies involving investigational concomitantly or within two weeks prior to entry into the study and during the course of the study

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Usual gluten-containing diet for healthy individuals | 1 month

SECONDARY OUTCOMES:
Usual gluten-free diet for celiac patients (home diet not modified for this trial) | 1 month

OTHER OUTCOMES:
Gluten-challenge in healthy individuals on GFD with 10 to 50 mg gluten | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Mª de Lourdes Moreno Amador, Dr, Study Chair — Department of Microbiology and Parasitology, University of Sevilla, Spain; Ángel Cebolla Ramírez, Dr, Study Chair — Biomedal S.L.; Ángeles Pizarro Moreno, Dr, Study Chair — Unidad Clínica de Aparato Digestivo, Hospital Universitario Virgen del Rocío, Sevilla, Spain; Alba Muñoz Suano, Dr, Study Chair — Biomedal, S.L., Sevilla, Spain; Isabel Comino Montilla, Dr, Study Chair — Department of Microbiology and Parasitology, University of Sevilla, Spain; Alfonso Rodríguez Herrera, Dr, Study Chair — Unidad de Gastroenterología y Nutrición, Instituto Hispalense de Pediatría. Sevilla, Spain; Francisco León, Dr, Study Chair — Celimmune, Bethesda, MD, USA; Carolina Carrillo Carrión, Study Chair — Biomedal, S.L., Sevilla, Spain; Carolina Sousa Martín, Professor, Principal Investigator — Department of Microbiology and Parasitology, University of Sevilla, Spain
Locations (1):
- Department of Microbiology and Parasitology, Faculty of Pharmacy, University of Seville, Seville, Seville, Spain

REFERENCES:
- [Background] Moron B, Bethune MT, Comino I, Manyani H, Ferragud M, Lopez MC, Cebolla A, Khosla C, Sousa C. Toward the assessment of food toxicity for celiac patients: characterization of monoclonal antibodies to a main immunogenic gluten peptide. PLoS One. 2008 May 28;3(5):e2294. doi: 10.1371/journal.pone.0002294. PMID 18509534
- [Background] Moron B, Cebolla A, Manyani H, Alvarez-Maqueda M, Megias M, Thomas Mdel C, Lopez MC, Sousa C. Sensitive detection of cereal fractions that are toxic to celiac disease patients by using monoclonal antibodies to a main immunogenic wheat peptide. Am J Clin Nutr. 2008 Feb;87(2):405-14. doi: 10.1093/ajcn/87.2.405. PMID 18258632
- [Background] Hausch F, Shan L, Santiago NA, Gray GM, Khosla C. Intestinal digestive resistance of immunodominant gliadin peptides. Am J Physiol Gastrointest Liver Physiol. 2002 Oct;283(4):G996-G1003. doi: 10.1152/ajpgi.00136.2002. PMID 12223360
- [Background] Shan L, Molberg O, Parrot I, Hausch F, Filiz F, Gray GM, Sollid LM, Khosla C. Structural basis for gluten intolerance in celiac sprue. Science. 2002 Sep 27;297(5590):2275-9. doi: 10.1126/science.1074129. PMID 12351792
- [Background] Comino I, Real A, Vivas S, Siglez MA, Caminero A, Nistal E, Casqueiro J, Rodriguez-Herrera A, Cebolla A, Sousa C. Monitoring of gluten-free diet compliance in celiac patients by assessment of gliadin 33-mer equivalent epitopes in feces. Am J Clin Nutr. 2012 Mar;95(3):670-7. doi: 10.3945/ajcn.111.026708. Epub 2012 Jan 18. PMID 22258271
- [Background] Comino I, Real A, Moreno Mde L, Montes R, Cebolla A, Sousa C. Immunological determination of gliadin 33-mer equivalent peptides in beers as a specific and practical analytical method to assess safety for celiac patients. J Sci Food Agric. 2013 Mar 15;93(4):933-43. doi: 10.1002/jsfa.5830. Epub 2012 Aug 6. PMID 22886585
- [Background] Real A, Comino I, Moreno Mde L, Lopez-Casado MA, Lorite P, Torres MI, Cebolla A, Sousa C. Identification and in vitro reactivity of celiac immunoactive peptides in an apparent gluten-free beer. PLoS One. 2014 Jun 25;9(6):e100917. doi: 10.1371/journal.pone.0100917. eCollection 2014. PMID 24963630
- [Derived] Moreno ML, Cebolla A, Munoz-Suano A, Carrillo-Carrion C, Comino I, Pizarro A, Leon F, Rodriguez-Herrera A, Sousa C. Detection of gluten immunogenic peptides in the urine of patients with coeliac disease reveals transgressions in the gluten-free diet and incomplete mucosal healing. Gut. 2017 Feb;66(2):250-257. doi: 10.1136/gutjnl-2015-310148. Epub 2015 Nov 25. PMID 26608460